CLINICAL TRIAL: NCT01463111
Title: Decision-Making in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Boadie W. Dunlop, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00050442; BDDM (Other: Other)
Record Dates: First submitted 2011-06-02; First posted 2011-11-01 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Manic depression; Mood stabilizer; Decision; Neuroeconomics
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Valproic Acid; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mood stabilizer (Other): Participants diagnosed with Bipolar Disorder will receive standard of care open-label treatment with a mood stabilizer for six weeks.
  Interventions: Drug: Lithium; Drug: Valproate; Drug: Lamotrigine

INTERVENTIONS:
Drug: Lithium — Open label treatment per standard of care for bipolar disorder for six weeks.
  Other Names: Eskalith
Drug: Valproate — Open label treatment per standard of care for bipolar disorder for six weeks.
  Other Names: Valproic Acid; Depakote
Drug: Lamotrigine — Open label treatment per standard of care for bipolar disorder for six weeks.
  Other Names: Lamictal

SUMMARY:
Forty subjects with bipolar disorder who are not receiving a mood-stabilizing medication for the treatment of their illness will participate in this study. The study aims to evaluate how decision-making is affected by treatment for bipolar disorder. Prior to beginning treatment, patients will complete questionnaires and a one-hour computer-administered assessment of decision-making. Differences between pre-post decision-making outcomes will be evaluated to examine whether the neuroeconomic concepts of risk aversion, loss aversion, risk tolerance and delay discounting are affected by treatment.

The overall goal of this study will be to identify whether decision-making in people with bipolar disorder is affected by treatment. Specifically the investigators will compare decision-making characteristics among bipolar patients prior to treatment with how these decision-making characteristics change over the course of 6 weeks of standard medication therapy for bipolar disorder. A total of 6 decision-making tasks and one control task will be administered via computer to eligible subjects. The investigators will evaluate decision-making under varying conditions of reward, risk, and uncertainty and over time. The investigators hypothesize that decision-making will improve across these assessments after 6 weeks of treatment.

DETAILED DESCRIPTION:
Participation in this study will require three study visits over 6 weeks. Subjects will be evaluated with the Structured Diagnostic Interview for DSM-IV to confirm diagnosis. They will also be administered the Hamilton Anxiety and Depression Rating Scales. Eligible subjects will then complete questionnaires related to their symptoms as well as decision-making and risk-taking, including: the Barratt Impulsiveness Scale, the Spielberger State-Trait Anxiety Inventory, and the Flinders Decision-making questionnaire. The Montgomery-Asburg Depression Severity scale to assess changes in depression symptom severity and the Young Mania Rating Scale to assess changes in manic symptom severity, will be conducted at screening, baseline, and endpoint. Patients will also be given the Childhood Trauma Questionnaire at baseline visit, to assess for a history of childhood trauma. The subjects will then complete the computer-generated decision-making tasks. Upon completion, the study physician will initiate standard-of-care treatment with a mood stabilizer (either lithium, valproate, or lamotrigine). Standard-of-care laboratory testing and psychiatric follow-up will be performed during the patient's study participation. After six weeks of treatment with a mood stabilizer, patients will again complete the decision-making computerized assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-65
2. Primary DSM-IV TR Diagnosis of Bipolar Disorder, type I, II or NOS.
3. Ability to visually read and understand English language
4. Not currently taking any mood stabilizer or antipsychotic medication.
5. Women of reproductive potential must be willing to take a medically approved form of birth control throughout the duration of the study.

Exclusion Criteria:

1. Meet criteria for substance abuse or dependence within three months of the screening visit.
2. Presents with a clinically significant suicide risk, as assessed by a study physician.
3. Presence of any unstable or central nervous system-related medical illness that would interfere with cognition or participation.
4. Women who are currently pregnant or lactating, or plan to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boadie W Dunlop, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Mood and Anxiety Disorders Program, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2011 through April 2016.
Pre-assignment Details: Of the 37 participants who consented for participation, 26 began study treatment. Eleven participants were screen failures.
Groups:
- Mood Stabilizer: Participants diagnosed with Bipolar Disorder received open-label treatment with a mood stabilizer for six weeks.
  Lithium, valproate, lamotrigine: Open label treatment per standard of care for bipolar disorder for six weeks.
Period: Overall Study
Arm/Group | Mood Stabilizer
Started | 26
Completed | 17
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mood Stabilizer
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.19 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14
  Other | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Vigilance Assessed by the Melbourne Decision Making Questionnaire (MDMQ)
Description: The MDMQ is a 22-item self report form assessing four different styles of decision making. Vigilance is considered the healthy, adaptive, decision-making style, reflecting consideration of an array of outcomes and ultimately rational decision-making. Scores range from 0-12. A higher score indicates that vigilance is used more frequently during decision making. A higher score indicates healthier decision making.
Time Frame: Baseline, Week 6
Population: Data was analyzed for participants who completed all study visits. Means are age-adjusted.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mood Stabilizer
Number analyzed (Participants) | 17
units on a scale | .176 (.778)

2. Primary Outcome: Change in Hypervigilance Assessed by the Melbourne Decision Making Questionnaire (MDMQ)
Description: The MDMQ is a 22-item self report form assessing four different styles of decision making. Hypervigilance is marked by hurried, anxious decision-making. Scores range from 0-10. A higher score indicates a "worse" score and that a hyper-vigilant decision making style is used more frequently.
Time Frame: Baseline, Week 6
Population: Data was analyzed for participants who completed all study visits. Means are age-adjusted.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mood Stabilizer
Number analyzed (Participants) | 17
units on a scale | -3.41 (3.08)

3. Primary Outcome: Change in Buckpassing Assessed by the Melbourne Decision Making Questionnaire (MDMQ)
Description: The MDMQ is a 22-item self report form assessing four different styles of decision making. The buckpassing decision-making style represents a tendency to leave decisions to others. Scores range from 0-12. A higher score indicates that the buckpassing decision-making style is used more frequently and represents a "worse" score.
Time Frame: Baseline, Week 6
Population: Data was analyzed for participants who completed all study visits. Means are age-adjusted.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mood Stabilizer
Number analyzed (Participants) | 17
units on a scale | -2.23 (3.72)

4. Primary Outcome: Change in Procrastination Assessed by the Melbourne Decision Making Questionnaire (MDMQ)
Description: The MDMQ is a 22-item self report form assessing four different styles of decision making. The procrastination decision-making style involves putting off making decisions. Scores range from 0-10. A higher score indicates that the procrastination decision-making style is used more and is considered a "worse" score.
Time Frame: Baseline, Week 6
Population: Data was analyzed for participants who completed all study visits. Means are age-adjusted.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mood Stabilizer
Number analyzed (Participants) | 17
units on a scale | 2.47 (3.41)

5. Secondary Outcome: Mean Difference in Barratt Impulsiveness Scale, Version 11 (BIS-11) Score
Description: The BIS-11 is a 30 item self-report questionnaire, used to assess three factors of impulsivity: 1). attentional impulsiveness, reflecting a difficulty concentrating or tolerating cognitive complexity, 2). motor impulsiveness, reflecting a tendency to act before thinking, and 3). non-planing impulsiveness, reflecting a lack of forethought about potential consequences. Items are scored on a 4-point scale: Rarely/Never = 1 Occasionally = 2 Often = 3 Almost Always/Always = 4. Attentional impulsivity scores range from 8-32. Motor impulsivity scores range from 11-44. Non-planning impulsivity scores range from 11-44. Total BIS-11 scores range from 30-120. A higher score reflects higher impulsivity across all sub-types.
Time Frame: Baseline, Week 6
Population: Data was analyzed for participants who completed all study visits. Means are age-adjusted.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mood Stabilizer
Number analyzed (Participants) | 17
units on a scale
  Attentional | -3.941 (3.716)
  Motor | -4.063 (3.108)
  Non-planning | -2.625 (5.227)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study.
Arm/Group | Mood Stabilizer
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 8/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mood Stabilizer (N=26)
Bartholin Cyst Removal (Surgical and medical procedures) | 1 (1)
Chlamydia Infection (Reproductive system and breast disorders) | 1 (1)
Hand Tremor (Nervous system disorders) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 2 (2)
Headache (Vascular disorders) | 6 (6)
Self-Injury (Psychiatric disorders) | 1 (1) — Self-injury refers to cutting oneself due to psychological reasons.
Nausea/Vomiting (Gastrointestinal disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Increased Urination (Renal and urinary disorders) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomach Ulcer (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Laryngitis (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Sedation (Psychiatric disorders) | 2 (2)
Thirst (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Weight Gain (Investigations) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Edema (General disorders) | 1 (1)
Impaired Concentration (Psychiatric disorders) | 1 (1)
Increased Sexual Interest (Psychiatric disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated Mood (Psychiatric disorders) | 1 (1)
Increased Anxiety (Psychiatric disorders) | 1 (1)
Dizziness/Vertigo (Ear and labyrinth disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes